CLINICAL TRIAL: NCT02432833
Title: Multicentre, Open Label, Randomized, Two-arm, Parallel-group Study to Assess Efficacy and Safety of ENVARSUS® Compared With Tacrolimus Used as Per Current Clinical Practice in the Initial Maintenance Setting in de Novo Kidney Transplant Patients
Acronym: STEADY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-06235AA1-01; 2014-004314-29 (EudraCT Number)
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Envarsus® (tacrolimus) (Experimental): prolonged-release tablets once daily and orally
  Interventions: Drug: ENVARSUS®
- Prograf or Advagraf (Active Comparator): Prograf® hard capsules, twice daily, oral formulation or Advagraf® prolonged-release hard capsules, once daily, oral formulation
  Interventions: Drug: PROGRAF®; Drug: ADVAGRAF®

INTERVENTIONS:
Drug: ENVARSUS® — Envarsus® tablets, once daily, oral formulation. Prolonged -release formulation of tacrolimus
  Arms: Envarsus® (tacrolimus)
Drug: PROGRAF® — Prograf® hard capsules, twice daily, oral formulation
  Arms: Prograf or Advagraf
Drug: ADVAGRAF® — Advagraf® prolonged-release hard capsules, once daily, oral formulation
  Arms: Prograf or Advagraf

SUMMARY:
The purpose of the study is to compare tacrolimus dosing of the new Envarsus®-based immunosuppressive regimen with current clinical practice (Prograf or Advagraf) over 6 months following de novo renal transplantation in a real-life setting in different European Countries.

DETAILED DESCRIPTION:
This is a Multicentre, Open label, Randomized, Two-arm, parallel-group study to assess efficacy and safety of Envarsus® compared with tacrolimus used as per current clinical practice in the initial maintenance setting in de novo kidney transplant patients. The study will be conducted in approximately 10 european countries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's signed informed consent obtained prior to any study-related procedure;
2. Adult men and women at least 18 years of age with end-stage renal disease who are recipients (or will be recipients) of a kidney transplant from a living or deceased donor;
3. No known contraindications to the administration of tacrolimus, other macrolides and study drugs excipients;
4. Patients must agree to use a highly reliable method of birth control;
5. Donor-recipient negative cross match test, and compatible AB0 blood type;
6. Able to swallow tablets and capsules

Exclusion Criteria:

1. Recipient of any transplanted organ other than kidney;
2. Recipient of a previous renal transplant;
3. Recipient of a kidney from a donor after cardiac death;
4. Recipient of a kidney from an AB0 incompatible or positive cross-match donor;
5. Current (not older than 3 months) anti-HLA Panel Reactive Antibody (PRA) levels higher than 30%. Whenever PRA, either complement-dependent cytotoxicity-PRA or calculated PRA , is not available, patients who are positive on solid-phase screening assay for anti-HLA antibodies must not be enrolled;
6. Recipient of a kidney with a cold ischemia time of ≥ 30 hours;
7. White blood cells count ≤ 2.8x109 cells/L unless ANC >1.0x109/L;
8. Platelet count < 50 x109 cells/L;
9. ALT or AST levels >3 times the normal upper limit during the 30 days prior transplant procedure;
10. Current abuse of drugs or alcohol;
11. Incapable of understanding purpose and risk of study, unable to give written informed consent or unwilling to comply with study protocol;
12. Treatment with any other investigational agent in the 30 days prior to enrolment;
13. Kidney recipients and/or donors positive for HCV (HCV-RNA positive or HCV-Ab positive respectively);
14. Kidney recipients and/or donors positive for HBV (HBV-DNA or HBS-Ag positive);
15. Recipients positive for HIV;
16. Patient or donor with current diagnosis or history of malignancy within the past 5 years except basal or non-metastatic squamous cell carcinoma of the skin successfully treated;
17. Uncontrolled concomitant infection, systemic infection requiring treatment or any other unstable condition that could interfere with study objectives;
18. Severe diarrhoea, vomiting, active peptic ulcer or GI disorder that may affect absorption of tacrolimus;
19. Known hypersensitivity to tacrolimus other macrolides and study drugs excipients;
20. Pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS are willing to use reliable methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Tacrolimus total daily dose (TDD) from week 3 to month 6 | from week 3 to month 6

SECONDARY OUTCOMES:
Tacrolimus blood trough level (TL). | from screening to months 6
number of dose adjustment | from screening to months 6
Occurrence of treatment failure | from screening to months 6
Delayed graft function | from screening to months 6
Acute rejection requiring treatment | from screening to months 6
Consumption of concomitant immunosuppressant medications | from screening to months 6
Treatment discontinuation | from screening to months 6

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, MD, Principal Investigator — Berlin, Germany
Locations (1):
- Chiesi farmaceutici Spa, Parma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Budde K, Rostaing L, Maggiore U, Piotti G, Surace D, Geraci S, Procaccianti C, Nicolini G, Witzke O, Kamar N, Albano L, Buchler M, Pascual J, Gutierrez-Dalmau A, Kuypers D, Wekerle T, Glyda M, Carmellini M, Tisone G, Midtvedt K, Wennberg L, Grinyo JM. Prolonged-Release Once-Daily Formulation of Tacrolimus Versus Standard-of-Care Tacrolimus in de novo Kidney Transplant Patients Across Europe. Transpl Int. 2022 Mar 21;35:10225. doi: 10.3389/ti.2021.10225. eCollection 2022. PMID 36017158
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-004314-29/results